CLINICAL TRIAL: NCT06774963
Title: A Phase 1, Open-label, Dose Escalation and Dose Expansion Study for LNCB74, a B7-H4 Targeted Antibody Drug Conjugate, as Monotherapy in Participants With Advanced Solid Tumors
Brief Title: A Phase 1 Study of LNCB74 in Advanced Solid Tumors
Acronym: LNCB74-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NextCure, Inc. (Industry)
Collaborators: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LNCB74-01; 168703 (Other: NextCure, Inc.)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Breast Cancer; Endometrial Cancer; Biliary Tract Cancer; Non-Small Cell Lung Cancer; Advanced or Metastatic Solid Tumors
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Biliary Tract Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 - Dose Escalation and Backfills (Experimental): Aim: Doses of LNCB74 will be escalated to determine the maximum tolerated dose (MTD), maximum administered dose (MAD) and/or recommended Phase 2 dose (RP2D). One or more dose levels will be backfilled for safety and additional biomarker data.
  Interventions: Drug: LNCB74
- Part 2 - Dose Expansion / Optimization (Experimental): Aim: The objectives of the Part 2 Dose Expansion/Optimization are: i) to evaluate safety, tolerability, anti-tumor activity, and pharmacodynamics of LNCB74 in a more homogenous population and ii) characterize the minimally safe and effective dose in a particular tumor type and determine recommended Phase 2 dose(s) (RP2D).
  Interventions: Drug: LNCB74

INTERVENTIONS:
Drug: LNCB74 — LNCB74 is an antibody drug conjugate being evaluated as a potential treatment for participants with advanced solid tumors. Participants will receive LNCB74 into the vein (IV; intravenously) in 21-day dosing cycles. Participants will continue treatment in the absence of unacceptable toxicities and unequivocal disease progression.

SUMMARY:
This is an open-label, phase 1, dose escalation and dose expansion study to determine safety and tolerability, and to determine the maximum tolerated dose and / or recommended phase 2 dose of LNCB74 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The participant provides written informed consent
2. ≥ 18 years of age on day of signing informed consent.
3. Participant with histologically or cytologically confirmed diagnosis of advanced unresectable and/or metastatic solid tumors
4. A male participant must agree to use contraception and refrain from sperm donation or expecting to father a child
5. A female participant is eligible to participate if she is not pregnant, not breastfeeding, not a woman of childbearing potential
6. Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology
7. Able to provide tumor tissue sample.
8. Willing to undergo fresh tumor biopsy at Screening and On-treatment if archival tissue not available
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
10. Life expectancy greater than or equal to 12 weeks as judged by the Investigator.
11. Have adequate organ function

Exclusion Criteria:

1. A WOCBP who has a positive serum pregnancy test (within 72 hours) prior to treatment.
2. Has received prior investigational agents within 4 weeks prior to treatment.
3. Has received anti-cancer chemotherapy (Immunotherapy (non-antibody-based therapy), retinoid therapy, hormonal therapy within 2 weeks prior to treatment.
4. Has received antibody-based anti-cancer therapy within 4 weeks prior to treatment.
5. Has received targeted agents and small molecules within 2 weeks or 5 half-lives, whichever is longer.
6. Has received prior platinum-based chemotherapy and progressed within 4 weeks of initiating therapy (platinum-refractory disease)
7. Has received an ADC with MMAE payload.
8. Has received prior radiotherapy within 2 weeks of start of study treatment for focal radiation or within 4 weeks for wide-field radiotherapy
9. Has received G-CSF or GM-CSF within 7 days prior to start of study treatment.
10. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
12. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
13. Has known active CNS metastases and/or carcinomatous meningitis
14. Has severe hypersensitivity (≥ Grade 3), known allergy or reaction LNCB74 or any of its excipients.
15. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
16. Has active ≥Grade 2 sensory or motor neuropathy.
17. Has active or chronic corneal disorders, other active ocular conditions requiring ongoing therapy or any clinically significant corneal disease.
18. Has an active infection requiring systemic therapy.
19. Any major surgery within 4 weeks of study drug administration.
20. Toxicity (except for alopecia) related to prior anti-cancer therapy and/or surgery, unless the toxicity is either resolved, returned to baseline or Grade 1, or deemed irreversible.
21. Prior organ or tissue allograft.
22. Uncontrolled or significant cardiovascular disease
23. Participants with serious or uncontrolled medical disorders.
24. Participants who are on total parenteral nutrition (TPN)
25. Participants with history of bowel obstruction within one month of screening
26. Participants with history of significant ascites requiring paracentesis within 2 weeks of screening
27. Has a known history of human immunodeficiency virus (HIV) infection with an acquired immune deficiency syndrome (AIDS)-defining opportunistic infection within the last year, or a current CD4 count <350 cells/µl
28. Has known active Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
29. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study
30. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 145 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of LNCB74 | 24 months
  Incidence of AEs, SAEs, AEs meeting protocol defined DLT criteria, AEs leading to discontinuation and death, and laboratory abnormalities per NCI CTCAE v5.0
Define a recommended Phase 2 dose (RP2D) of LNCB74 | Up to 24 months
  Maximum tolerated dose (MTD), maximum administered dose (MAD) and/or recommended Phase 2 dose (RP2D) of LNCB74

SECONDARY OUTCOMES:
Characterize the immunogenicity of LNCB74 | 24 months
  Incidence of anti-drug antibodies to LNCB74
Objective Response Rate (ORR) | 24 months
  Objective Response Rate (ORR) per RECIST v1.1
Duration of Response (DOR) | 24 months
  Duration of response per RECIST v1.1
Disease Control Rate (DCR) | 24 months
  Disease control rate per RECIST v1.1
Progression Free Survival Rate (PFSR) | 6 months
  Progression Free Survival Rate per RECIST v1.1
Correlate B7-H4 Expression with Objective Response Rate (ORR) | 24 months
  To determine B7-H4 expression by immunohistochemistry in a central lab and correlate B7-H4 expression with Objective Response Rate (ORR)
Correlate B7-H4 Expression with Duration of Response (DOR) | 24 months
  To determine B7-H4 expression by immunohistochemistry in a central lab and correlate B7-H4 expression with Duration of Response (DOR)
Correlate B7-H4 Expression with Disease Control Rate (DCR) | 24 months
  To determine B7-H4 expression by immunohistochemistry in a central lab and correlate B7-H4 expression with Disease Control Rate (DCR)
Correlate B7-H4 Expression with Progression Free Survival (PFS) | 24 months
  To determine B7-H4 expression by immunohistochemistry in a central lab and correlate B7-H4 expression with Progression Free Survival (PFS)
Progression Free Survival (PFS) | 24 months
  Progression Free Survival per RECIST v1.1
Time to Peak Drug Concentration (Tmax) of LNCB74 | Cycle 1 Days 1, 3, 8 and 15; Cycle 3 Days 1, 3, 8 and 15; Day 1 of Cycles 2, 4, 5, 7 and 9
  To evaluate the Time to Peak Drug Concentration (Tmax) of LNCB74
Area Under the Curve (AUC) of LNCB74 | Cycle 1 Days 1, 3, 8 and 15; Cycle 3 Days 1, 3, 8 and 15; Day 1 of Cycles 2, 4, 5, 7 and 9
  To evaluate the Area Under the Curve (AUC) of LNCB74
Half-life (T1/2) of LNCB74 | Cycle 1 Days 1, 3, 8 and 15; Cycle 3 Days 1, 3, 8 and 15; Day 1 of Cycles 2, 4, 5, 7 and 9
  To evaluate the Half-life (T1/2) of LNCB74
Maximum Serum Concentration (Cmax) of LNCB74 | Cycle 1 Days 1, 3, 8 and 15; Cycle 3 Days 1, 3, 8 and 15; Day 1 of Cycles 2, 4, 5, 7 and 9
  To evaluate the Maximum Serum Concentration (Cmax) of LNCB74

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Hoag Family Cancer Institute, Newport Beach, California
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Ctr at Hackensack Univ. Med Ctr., Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Sidney Kimmel Comprehensive Center at Jefferson, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - MD Anderson, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - UT Health San Antonio - MD Anderson Cancer Center, San Antonio, Texas
  - Intermountain/LDS Hospital Ph 1 Research Program, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No